CLINICAL TRIAL: NCT07082777
Title: Recovery in Telling Life Stories (RETELL): Testing a Narrative Identity Intervention for Personal Recovery in Individuals With Severe Mental Illness
Brief Title: Recovery in Telling Life Stories
Acronym: RETELL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Dinne Christensen, Principal Investigator ,Postdoc, PhD, University of Aarhus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0367531, 3878; 1-10-72-56-25 (Other: VEK Region Midt)
Record Dates: First submitted 2025-07-04; First posted 2025-07-24 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia Disorders; Personality Disorders; Obsessive - Compulsive Disorder; Anxiety Disorders; Recurrent Depressive Disorder; PTSD - Post Traumatic Stress Disorder; Hyperkinetic Disorders; Eating Disorders; Bipolar Disorders; Aspergers Syndrome
Keywords: personal recovery; recovery; narrative identity; narrative therapy; severe mental illness
MeSH Terms: conditions — Schizophrenia; Personality Disorders; Compulsive Personality Disorder; Anxiety Disorders; Depressive Disorder; Combat Disorders; Attention Deficit Disorder with Hyperactivity; Feeding and Eating Disorders; Bipolar Disorder; Asperger Syndrome; Mental Disorders | interventions — Narrative Therapy; Salvage Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RETELL (Experimental): Narrative therapy to support personal recovery, delivered individually over 8-12 sessions.
  Interventions: Behavioral: Narrative therapy

INTERVENTIONS:
Behavioral: Narrative therapy — The intervention is structured around 4 central tasks focusing on different aspects of narrative repair. Task 1: Introduction to life story exploration and building alliance. Task 2: Explore and process the impact of mental illness on identity, externalizing negative narratives, and making sense of emotional responses such as guilt, grief, or shame. Task 3: Identify positive identity conclusions (e.g., strengths, values, skills) from past or current life experiences, and support their integration into the personal narrative. Task 4: Support the imagining of a realistic and hopeful future narrative, grounded in insights of previous sessions. Tasks 1-4 are addressed in a total of 8-12 sessions, depending on the specific user needs. Sessions will have an app. duration of 45-60 mins and will be delivered by the PI who is a trained therapist and psychologist (MSc. Psych.), receiving ongoing supervision. The intervention manual will be made freely available in relation to study publication.
  Other Names: Recovery in Telling Life Stories (RETELL)

SUMMARY:
This project tests the Recovery In Telling Life Stories (RETELL) intervention, aimed at supporting personal recovery in people with severe mental illness (SMI). While many of those with SMI experience symptom control, their quality of life often remains low due to social loss, negative self-perceptions, and identity-related challenges not addressed by standard treatments. Through a process of narrative repair, the RETELL intervention helps participants explore the personal consequences of mental illness while supporting the enhancement of narratives that strengthen identity and foster well-being. The intervention is delivered across 8-12 sessions and will be assessed for feasibility of both the intervention and study procedures. We will also explore its preliminary impact on recovery, quality of life, symptoms, functioning, self-stigma, and personality, using a multiple single-case A-B-A design. We expect the intervention and study procedures to show acceptable feasibility. We further hypothesize that participants' scores on recovery and well-being will be low at baseline, improve during the intervention, and remain higher after the intervention ends and at 3-month follow-up. This study will provide a foundation for future randomized controlled trials.

DETAILED DESCRIPTION:
This project tests the Recovery In Telling Life Stories (RETELL) intervention, an intervention developed to support personal recovery in individuals with severe mental illness (SMI).

Research shows that many people with SMI experience low quality of life even when their symptoms are in remission and functional level, e.g. cognitive remediation. This is not only due to the illness itself but also to the consequences that often accompany it, such as the loss of social and occupational roles and the development of negative self-perceptions. These challenges are only to a limited extent addressed by existing treatments, which typically focus on symptom reduction.

Personal recovery is about living a satisfying and meaningful life despite the potential constraints associated with mental illness. A major barrier to this process can arise when a person develops an understanding of themself (a narrative identity) characterized by shame, low self-esteem, and self-stigmatization. When negative identity conclusions dominate, it can be difficult to experience well-being, meaning in life, or hope for the future.

Despite an increasing focus on personal recovery in mental health care systems globally, evidence-based methods to support the recovery process are limited. In this project, we develop and test the RETELL intervention, designed to support personal recovery by helping participants process the personal consequences of mental illness and identify and cultivate positive identity conclusions and personal strengths. In RETELL, the participants are guided through this process, which we refer to as narrative repair, over a structured sequence of 8-12 sessions. Across these sessions, participants are guided in telling their life story and in constructing preferred and empowering narratives about themselves and their future.

The intervention will be tested in a mixed methods study using a one-arm multiple single-case intervention design with an A-B-A structure. This includes a pre-intervention phase (T1) with four weeks of outcome measurements, an intervention phase (T2) continuing with the same measures every second week, 4 weeks of post-intervention measurements (T3), and 4 weeks of follow-up measurements starting 3 months after intervention completion (T4). Data will be collected in electronic surveys and qualitative interviews. The primary aim is to assess intervention feasibility including potential to improve recovery and quality of life. It is aimed to recruit 20 participants diagnosed with SMI within the timeframe allowed by the study plan.

Feasibility will be assessed in terms of both intervention and study procedure feasibility, as this study will form the basis for larger randomized controlled trials. Intervention feasibility will be evaluated based on treatment dropout, treatment satisfaction and trajectory of self-reported recovery compared to pre-intervention. Feasibility will be indicated by < 30% dropout, a mean sum score of ≥ 20 on the Client Satisfaction Questionnaire, and increase or stability of self-reported recovery throughout the study period compared to pre-intervention. Study procedure feasibility includes recruitment acceptance rate, questionnaire response rate and study dropout rate. We tentatively propose a ≥ 50% recruitment acceptance rate, ≥ 75% questionnaire response rate and ≤ 25% study dropout rate as indicating acceptable study feasibility.

Secondary outcomes include well-being, domain-specific recovery, overall functioning, symptom levels, and self-stigmatization. In addition, changes from pre- to post-intervention in personality trait scores will be explored. Statistical analyses will include dependent t-tests to examine effect sizes and changes in quantitative outcomes, and these will be interpreted with attention to clinical significance. Finally, interviews about participants' experiences with the intervention will be thematically analyzed to identify perceived helpful elements, potential mechanisms of change and to inform the refinement of the programme theory.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18 and 65 years
* A self-reported principal diagnosis of one or more of the following: schizophrenia (F20), bipolar disorder (F31), personality disorders (F60), obsessive-compulsive disorder (F42), anxiety disorders (F41), recurrent depressive disorder (F33), eating disorders (F50), hyperkinetic disorders (F90), post-traumatic stress disorder (F43.1), Asperger syndrome (F84.5)
* Not in full recovery (Brief INSPIRE-O < 50)
* Danish language proficiency
* Medication stabilized (i.e., same type and dosage for a minimum of 8 weeks)
* Ability and willingness to give informed consent

Exclusion Criteria:

* Self-reported diagnosis of mental retardation (F70-79) and/or organic mental disorder (F00-09)
* Psychiatric symptoms, thoughts of self-harm and/or substance abuse of self-reported severity which are likely to prevent one or all of the following: attendance at scheduled sessions, completion of questionnaires before, during and after the intervention, meaningful engagement in the therapeutic process
* Psychiatric hospitalization in the past 4 weeks
* Prior conviction of violent crime
* Currently homeless
* Currently in psychotherapy initiated within the past 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Intervention feasibility: Treatment dropout rate | Through intervention phase (T2), between 8-12 weeks
  Treatment dropout is defined as participation in less than three out of the four therapeutic tasks of the intervention. Feasibility will be indicated by a dropout rate < 30%.
Intervention feasibility: Satisfaction with treatment (quantitative) | Post-intervention (T3)
  Participant-reported treatment satisfaction using the using the Client Satisfaction Questionnaire (CSQ), a brief, standardized self-report measure designed to assess clients' overall satisfaction with healthcare or psychological services. It consists of 8 items rated on a Likert scale, covering aspects such as service quality, perceived helpfulness, and whether the service met the client's needs. Total score range: 8-32, with higher numbers indicating greater satisfaction. Feasibility will be indicated by a mean score of 20 or above.
Intervention feasibility: Change from pre-intervention throughout the intervention to post-intervention and follow-up in personal recovery | Pre-intervention (T1), intervention (T2), post-intervention (T3) and follow-up (T4)
  Recovery will be assessed using the Brief INSPIRE-O, consisting of 5 items reflecting five dimensions of personal recovery: connectedness with others, hope and optimism for the future, positive identity, meaning in life, and empowerment, with a score range of 0-100. Feasibility will be indicated by stability or increase throughout the study period compared to pre-intervention.

SECONDARY OUTCOMES:
Intervention feasibility: Number of participants with treatment-related adverse events | From the beginning of the intervention (T2) to the final 3-month follow-up (T4)
  Self-reported adverse events will be monitored during the intervention phase (T2) by systematic inquiry to hospitalization, thoughts of self-harm and suicide attempts, as well as at follow-up points (T3 and T4) by use of the DSM-5-TR Self-Rated Level 1 Cross-Cutting Symptom Measure for Adults. Participants will also have the opportunity to anonymously report adverse events to a project staff member.
Intervention feasibility: Satisfaction with the therapeutic alliance | Intervention phase (T2)
  Participant-reported quality of the therapeutic alliance using the Session Rating Scale (SRS), a visual analogue scale (ranging from 0 to 10) that allows individuals to provide feedback on key aspects of the session, such as the therapeutic alliance and overall experience.
Intervention feasibility: Satisfaction with treatment (qualitative) | Post-intervention (T3)
  Participant-reported treatment satisfaction in qualitative, semi-structured interviews
Change from pre-intervention throughout the intervention to post-intervention and follow-up in well-being | Pre-intervention (T1), intervention (T2), post-intervention (T3) and follow-up (T4)
  Well-being will be assessed using the 5-item World Health Organization's Well-Being Index (WHO-5), designed to measure subjective well-being. Score range: 0-100.
Change from pre-intervention to post-intervention and follow-up in domain-specific recovery | Pre-intervention (T1), post-intervention (T3) and follow-up (T4)
  Domain-specific recovery will be assessed using the Recovery Assessment Scale-Domains and Stages (RAS-DS), a self-report measure designed to capture an individual's subjective experience of recovery across multiple life domains. The scale assesses four key domains: Doing Things I Value, Looking Forward, Mastering My Illness, and Connecting and Belonging, each reflecting different aspects of personal recovery. Items are rated on a 4-point Likert scale, ranging from 1 (Untrue) to 4 (Completely true). The total scale score ranges from 38-152, with higher scores indicating greater perceived recovery. The RAS-DS is grounded in a consumer-oriented understanding of recovery and has demonstrated good psychometric properties across various mental health populations.
Change from pre-intervention to post-intervention and follow-up in functioning and disability | Pre-intervention (T1), post-intervention (T3) and follow-up (T4)
  Functioning and disability will be assessed using the World Health Organization Disability Assessment Schedule 2.0 (WHODAS) 12-item version, a brief, standardized self-report instrument developed to assess difficulties in daily functioning across the past 30 days. Responses are scored on a 5 point Likert scale: None (0), Mild (1), Moderate (2), Severe (3), and Extreme/Cannot Do (4).
Change from pre-intervention to post-intervention and follow-up in symptomatic status | Pre-intervention (T1), post-intervention (T3) and follow-up (T4)
  Symptomatic status will be assessed using the DSM-5-TR Self-Rated Level 1 Cross-Cutting Symptom Measure for Adults, a standardized screening tool to assess a broad range of psychiatric symptoms across multiple diagnostic domains. The measure includes 23 items covering 13 symptom domains (e.g., depression, anxiety, psychosis, sleep problems, and substance use), each rated on a 5-point scale from 0 (none) to 4 (severe), reflecting symptom severity over the past two weeks.
Change from pre-intervention to post-intervention and follow-up in self-stigmatization | Pre-intervention (T1), post-intervention (T3) and follow-up (T4)
  Self-stigmatization will be assessed using the 10-item version of the Internalized Stigma of Mental Illness Scale (ISMI), a brief, validated self-report measure used to assess the degree to which individuals internalize negative beliefs and stereotypes about mental illness across the following subscales: Alienation, Discrimination Experience, Social Withdrawal, Stereotype Endorsement, and Stigma Resistance. Responses are a 4-point Likert scale ranging from strongly disagree (1) to strongly agree (4) for a total score range of 10 to 40, with higher scores representing more severe internalized stigmatization.
Change from pre-intervention to follow-up in Big 5 personality traits | Pre-intervention (T1) and post-intervention (T3)
  Big 5 personality traits will be assessed using the Big Five Inventory-2-S (BFI-2-S), a 30-item short form of the BFI-2 designed to measure the five broad personality domains: Extraversion, Agreeableness, Conscientiousness Neuroticism, and Openness to Experience. Each trait is assessed with 6 items rated on a 5-point Likert scale ranging from 1 (disagree strongly) to 5 (agree strongly).
Study procedure feasibility: Acceptance rate | Study recruitment phase, approximately 15 months
  The proportion of participants enrolled from the number of individuals who received oral and written information about the study from the study coordinator, and were found to be eligble during screening.
Study procedure feasibility: Questionnaire response rate | Throughout study completion, an average of approximately 35 weeks.
  The average percentage of questionnaires completed within each batch (e.g., T1) and overall (T1-T4).
Study procedure feasibility: Study drop-out rate | Throughout study completion, an average of approximately 35 weeks.
  Rate of nonresponse to any complete batch of questionnaires during intervention phase, at postintervention or follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Dorthe K. Thomsen, PhD, Study Chair — University of Aarhus
Locations (1):
- Aarhus Univerity, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data from this study will not be shared due to their highly sensitive nature. The data include detailed narratives and information related to mental health, which pose a significant risk of re-identification-even if direct identifiers are removed. Given the ethical obligation to safeguard participants' privacy and the strict requirements of data protection regulations (e.g., GDPR), we have determined that sharing IPD would not be compatible with the informed consent provided by participants or with responsible research conduct. Therefore, only aggregate findings will be shared upon request, and only for research purposes.

REFERENCES:
- [Background] Thomsen, D. K., et al. (2023). Storying Mental Illness and Personal Recovery. Cambridge, Cambridge University Press.